CLINICAL TRIAL: NCT06190574
Title: Diagnostic Efficacy and Prognostic Value of 18F-FDG PET/CT (MR) in Pediatric Solid Blastoma
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: XLan-1218
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-12

CONDITIONS: 18F-FDG; Neuroblastoma; Hepatoblastoma; Wilms Tumor
MeSH Terms: conditions — Neuroblastoma; Hepatoblastoma; Wilms Tumor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Telephone follow-up — Telephone follow-up

SUMMARY:
the primary histologic origin of extracranial solid tumors in children is malignant embryonic cells, including Neuroblastoma (NB) , Hepatoblastoma(HB), and kidney, wilms' tumor(WT). Their main clinical symptoms are large abdominal masses, the most common lymph node metastasis . NB accounts for 15% of childhood cancer deaths, but some low-risk NB can disappear on its own. The International Neuroblastoma Risk Group Staging System (INRGSS) was used to determine Risk before NB treatment, whereas the INRGSS was entirely based on the Neuroblastoma diagnosis, illustrating the importance of imaging in the assessment of NB.18F-FDG is the most commonly used agent in PET imaging of tumor. It can reflect the glucose metabolism of tumor and is widely used in the diagnosis, staging, evaluation of curative effect and prognosis prediction of tumor In this study, the investigators retrospectively analyzed 18F-FDG PET/CT or PET/MRI images from patients with NB, HB, and WT. The investigators sought to assess whether these images provide useful information for diagnosis and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. age < 18 years,
2. have pathological results or definite clinical diagnosis as the gold standard.

Exclusion Criteria：

1. had surgery or chemotherapy before imaging,
2. accompanying other tumors,
3. diabetic patients or patients with fasting blood glucose ≥ 200 mg/dL.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: We reviewed the electronic medical record and imaging data of 47 children who underwent 18F- FDG PET/CT or PET/MR for the diagnosis of suspected NB, HB or WT from Jan 1, 2013, to Aug 30, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Region of Interest (ROI) | up to 2 years
  The presence of non-physiological uptake or uptake in a tissue structure can be considered pathological. The lesion intake is higher than the health organization and is classified as clearly positive. The lesion and the surrounding normal tissue ROI, measure the SUV, TLG and MTV.
Sensitivity and specificity of diagnosis and staging | up to 2 years
  Comparison of the high uptake portion of a pet image suspected to be a histiocytoma for consistency with pathological findings, using the pathological section as the gold standard to calculate the sensitivity and specificity of the diagnostic.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Principal Investigator — Study Principal Investigator Wuhan Union Hospital, China
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided